CLINICAL TRIAL: NCT01067924
Title: Motivational Interviewing to Promote Maintenance of Physical Activity in People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Marni Armstrong, PhD student, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22490
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes, motivational interviewing, physical activity maintenance, physical activity adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational interviewing (Experimental)
  Interventions: Behavioral: Motivational interviewing
- Standard of care (Active Comparator)
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing — Intervention arm will receive 2 motivational interviewing session aimed at increasing maintenance of physical activity upon the completion of a supervised exercise program. Motivational interviews will occur at the end of the structured program and at 3 months post program completion. Outcomes will be collected at 6 months post-program.

SUMMARY:
The purpose of the study is to assess the effectiveness of motivational interviewing in promoting maintenance of physical activity in people with Type 2 diabetes (T2D) upon the completion of a structured exercise program.

Participants with T2D who are new graduates of a supervised exercise program will be randomly assigned to either standard care (SC) or to standard care and in addition, participate in two individual motivational interview (MI) sessions (SC + MI).

The primary outcome will be change in physical activity behavior assessed by the Godin Leisure and Exercise questionnaire. Secondary outcomes will include change in blood glucose control (A1C), BMI, six minute walk-test, QoL, and self-efficacy.

Outcomes will be measured in groups at baseline, end of program, 3 months and 6 months post-program.

ELIGIBILITY:
Inclusion Criteria:

* a) self-reported physician diagnosed T2D, included are those who are treated with diet alone, oral medication and insulin
* b) clearance by Living Well clinical staff to exercise through GXT algorithm and triaged to "Keep Going" level class,
* c) at least 18 years of age,
* d) ability to read and write in English.

Exclusion Criteria:

* a) insulin therapy that began less than 2 years after T2D diagnosis,
* b) changes during the previous 2 months in oral hypoglycemic

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-09; Primary Completion 2012-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in physical activity as measured by the GODIN physical activity questionnaire | baseline, 3, 6 months post program

SECONDARY OUTCOMES:
Change in Hemoglobin A1C, BMI, six minute walk-test, QoL, and self-efficacy. | Baseline, 3, 6 months post-program

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Sigal, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada